CLINICAL TRIAL: NCT07276594
Title: The Effect of White Noise and Stress Balls Applied During NST to Pregnant Women Scheduled for Cesarean Section on Anxiety, Fetal Well-being, and Fear of Surgery
Brief Title: Impact of White Noise and Stress Balls on Anxiety, Fetal Well-Being, and Surgical Fear in Elective Cesareans
Acronym: Nonstrestest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, nurten özçalkap, Asistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/140
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Elective Cesarean Section; Non Stress Test (NST)
Keywords: Elective Cesarean Section,; anxiety,; fear of surgery,; fetal well-being; Non Stress Test
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This research was conducted with the randomized control group pretestposttest trial model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): only white noise group
  Interventions: Other: only white noise
- Group 3 (Experimental): white noise + stress ball group
  Interventions: Other: White noise + stress ball
- Group 2 (Experimental): Only stress ball
  Interventions: Other: only stress ball
- Group 4 (No Intervention): standard care group

INTERVENTIONS:
Other: only white noise — White noise listening intervention was initiated 15 minutes before the NST application. Both white noise listening and stress ball squeezing and releasing were performed throughout the NST application and for15 minutes after the application ended.
  Arms: Group 1
Other: only stress ball — The stress ball intervention was initiated 15 minutes before the NST application. Throughout the NST application and for 15 minutes after the application ended, the stress ball squeezing and releasing exercise was performed.
  Arms: Group 2
Other: White noise + stress ball — White noise + stress ball intervention, starting 15 minutes before the NST application, continuing throughout the NST application, and continuing for 15 minutes after the application ends, involving both listening to white noise and squeezing and releasing the stress ball.
  Arms: Group 3

SUMMARY:
This study aims to determine the effect of white noise and stress balls administered during NST on anxiety, fetal well-being, and fear of surgery in pregnant women scheduled for planned cesarean sections. A total of 168 pregnant women will be included in the study, divided into 4 groups (white noise group, stress ball group, white noise group + stress ball group, and control group).

DETAILED DESCRIPTION:
Participants will only be exposed to white noise and stress ball therapy; no invasive procedures will be performed.

Experimental Group Participants will be invited to participate in the study through face-to-face interviews conducted individually. Participants assigned to the experimental group via randomization will be informed about the study and their consent will be obtained.

Pregnant women who agree to participate in the study will receive the intervention starting 15 minutes before the NST application and continuing throughout the NST application; those in the white noise group will listen to white noise, those in the stress ball group will receive the stress ball intervention, and those in the white noise + stress ball group will listen to white noise and receive the stress ball intervention. Before the session begins, the "Informative Information Form," "NST Findings Record Form," "Surgical Fear Scale," and "Spielberger State Anxiety Inventory" will be administered. After the NST application, the "NST Findings Record Form," "Spielberger State Anxiety Inventory," and "Surgical Fear Scale" will be administered.

Control Group Participants will be invited to participate in the study through face-to-face interviews conducted individually. Participants in the control group will be informed about the study and their consent will be obtained according to the randomization method. No intervention other than routine care will be performed. Participants in the control group will first be administered the "Informative Information Form," "NST Findings Record Form," "Surgical Fear Scale," and "Spielberger State Anxiety Inventory" for the pre-test. After the NST application is completed, the "NST Findings Record Form," "Spielberger State Anxiety Inventory," and "Surgical Fear Scale" will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  * No communication barriers
  * 32-38 weeks of gestation,
  * Planning a cesarean delivery,
  * No risk factors during pregnancy (preeclampsia, IUGR, premature rupture of membranes, gestational diabetes, etc.),
  * Single pregnancy,
  * No health problems (such as fetal anomaly, intrauterine growth restriction) in the fetus

Exclusion Criteria:

* Having any risk factors during pregnancy (preeclampsia, IUGR, premature rupture of membranes, gestational diabetes, etc.)

  * Having a multiple pregnancy
  * Having a fetus with any health problems (such as fetal anomaly, intrauterine growth restriction) Exclusion criteria from the study
  * Incomplete responses to the survey questions
  * Wish to withdraw from the study,
  * Development of a risk condition during pregnancy,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women who will have a elective cesarean section
Enrollment: 168 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Surgical Fear Questionnaire (SFQ) | preoperative
  to determine the level of fear caused by the short- and long-term outcomes of surgical operations in patients undergoing elective surgery
Spielberger State Anxiety Inventory | preoperative
  to measure state anxiety levels in normal and abnormal individuals. It is a self-assessment type measure consisting of short statements. The State Anxiety Inventory was developed to measure a person's anxiety at a specific moment. The 20-item State Anxiety Inventory is a measure that determines how an individual feels at a specific moment and under specific conditions. The feelings or behaviors expressed in the items of the State Anxiety Inventory are answered by selecting one of the options (1) not at all, (2) a little, (3) very much, (4) completely) according to the degree of intensity. There are 10 reverse-scored items in the inventory. These items are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The state anxiety score is calculated by adding 50 points to the difference between the total weighted scores of the direct and reverse items.
Personal Information Form (PIF) | preoperative
  This form was developed by researchers to identify some of the individual characteristics of pregnant women. It includes questions about some of the women's sociodemographic characteristics (such as age, education level, income and employment status, surgical history, and history of cesarean section).
NST Finding Form The Non-Stress Test (NST) | preoperative
  It is an assessment method that measures the response of fetal heart rate to fetal movements over time. If at least two or more fetal movements are observed during a 20-minute monitoring period and an increase in heart rate of at least 15 beats (acceleration) lasting at least 15 seconds occurs during these movements, the result is considered reactive or "reassuring" (ACOG, 2019). Furthermore, the absence of decelerations on the NST and an average fetal heart rate between 110-160 bpm are indicators of a healthy fetal condition (Güngör, 2016; Nacar & Türkmen, 2022; Umana, 2022). In this context, the NST finding form was prepared by researchers, guided by the literature, to include the mean fetal heart rate, acceleration and deceleration status, and reactive/non-reactive status.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Özçalkap, Asistant Professor, Principal Investigator — inonü üniversity; Emel GÜÇLÜ CİHAN, Associate Professor, Study Chair — SÜTÇÜ İMAM UNIVERSTY; SEVDA TAŞTAN, Study Chair — Adiyaman University
Locations (4):
- Turkey (Türkiye) (4):
  - Adıyaman Üniversitesi, Adıyaman
  - Kahramanmaraş Sütçü İmam Üniversitesi, Kahramanmaraş
  - İnonu Universty, Malatya
  - İnonü Universty, Malatya

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Öner N, Le Compte A. Süreksiz Durumluk/Sürekli Kaygı Envanteri El Kitabı, 1. Baskı, Boğaziçi Üniversitesi Yayınları, İstanbul, 1983. ss: 1-26.